CLINICAL TRIAL: NCT05079685
Title: HyFoSy Versus HSG as a Diagnostic Technique for Tubal Patency: a Prospective Case-control Study.
Brief Title: HyFoSy Versus HSG as a Diagnostic Technique for Tubal Patency.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-HyF
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Tubal Patency; Sterility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases-Control: Women aged 18-39 years, with BMI <30 and good ovarian reserve, undergoing study for primary sterility, subsidiary of conducting tubal patency studies to rule out pathology of the same and thus be able to perform Spousal or Donor IA.

SUMMARY:
Observational, single-center, prospective case-control study, in which each patient is his own control.

It focuses on the study of tubal patency and establishing the agreement of results between HyFoSy and HSG.

DETAILED DESCRIPTION:
Observational, single-center, case-control study in which tubal pathology is studied in the context of a Basic Sterility Study.

The main objective of this study is to demonstrate the concordance of this new diagnostic test (HyFoSy) with HSG, which is the common technique to visualize tubal patency. Once demonstrated concordance, we also want to carry out a cost-effectiveness study and demonstrate through different scales the greater ease of the test, less time to perform and less pain for the patient.

It is a study in which the patients are women between 18-39 years old, undergoing study for primary sterility, with a BMI <30, AMH> 0.6 (good ovarian reserve).

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-39 years, under study for primary sterility, with BMI <30, AMH> 0.6 (good ovarian reserve), subsidiaries of Conjugal or Donor IA, according to the 2019 SAS Reproduction Guide.

Exclusion Criteria:

* Women <19 or> 39 years old, BMI> 30, secondary sterility, previous tubal sterilization, that is, the ART exclusion criteria according to the 2019 SAS Reproduction Guide.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — It is a study in which tubal patency is studied through the technique of visualization of the tubes. The patients in the study will be only women.
Study Population: Women aged 18-39 years, with BMI <30 and good ovarian reserve, undergoing study for primary sterility, subsidiary of conducting tubal patency studies to rule out pathology of the same and thus be able to perform Spousal or Donor IA.
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Study of tubal patency and establish the concordance of results between HyFoSy and HSG. | Up to 48 weeks.
  Concordance study between HyFoSy and HSG. It is a qualitative study (yes / no).

SECONDARY OUTCOMES:
Rate of occurrence of complications in the patients included in the study. | Up to 48 weeks.
  Expand the knowledge of the complications in the clinical practice of HyFoSy, confirming the lower perception of pain and the therapeutic effect of HyFoSy.
Time costs of performing HyFoSy versus HSG. | Up to 48 weeks.
  Compare the time it takes to see the effect of the study drug compared to HSG.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Morales Bueno, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen macarena, Seville, Spain